CLINICAL TRIAL: NCT05587374
Title: Cadonilimab as Induction-adjuvant PD-1/CTLA-4 Bispecific Blockade Combined With Induction Chenotherapy and Concurrent Chemoradiotherapy in High-risk Locoregionally-advanced Nasopharyngeal Carcinoma: a Multicenter, Randomized, Controlled, Multicenter, Phase 3 Clinical Trial
Brief Title: Cadonilimab (PD-1/CTLA-4 Bispecific Blockade) and Chemoradiotherapy in Nasopharyngeal Carcinoma (GEMSTONE)
Acronym: GEMSTONE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Akeso Pharmaceuticals, Inc. (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-019
Record Dates: First submitted 2022-10-18; First posted 2022-10-20 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Nasopharyngeal Carcinoma; Nasopharyngeal Cancer
Keywords: immunotherapy; PD-1/CTLA-4 Bi-specific Antibody; Chemoradiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Nasopharyngeal Neoplasms | interventions — Gemcitabine; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Masking Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cadonilimab arm (Experimental): Patients will receive induction chemotherapy with gemcitabine (1g/m2, d1 & 8 of every cycle) and cisplatin (80mg/m2, d1 of every cycle), every 3 weeks for 3 cycles before radiation. Definitive intensity-modulated radiotherapy (IMRT) of 6996cGy in 33 fractions will be given. Concurrent cisplatin of 100mg/m2 will be administered every 3 weeks for 2 cycles during IMRT. Cadonilimab 10mg/kg will be given every 3 weeks for 3 cycles in induction chemotherapy and for 14 cycles in adjuvant chemotherapy, started on day 1 of induction chemotherapy and adjuvant chemotherapy, respectively.
  Interventions: Drug: Cadonilimab; Drug: Gemcitabine; Drug: Cisplatin; Radiation: Intensity-modulated radiotherapy
- Chemoradiation arm (Active Comparator): Patients will receive induction chemotherapy with gemcitabine (1g/m2, d1 & 8 of every cycle) and cisplatin (80mg/m2, d1 of every cycle), every 3 weeks for 3 cycles before radiation. Definitive intensity-modulated radiotherapy (IMRT) of 6996cGy in 33 fractions will be given. Concurrent cisplatin of 100mg/m2 will be administered every 3 weeks for 2 cycles during IMRT.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Radiation: Intensity-modulated radiotherapy

INTERVENTIONS:
Drug: Cadonilimab — Cadonilimab 10mg/kg will be given every 3 weeks for 3 cycles in induction chemotherapy and for 14 cycles in adjuvant chemotherapy, started on day 1 of induction chemotherapy and adjuvant chemotherapy, respectively.
  Other Names: PD-1/CTLA-4 bi-specific antibody
  Arms: Cadonilimab arm
Drug: Gemcitabine — Gemcitabine 1g/m2, d1 & 8 of every cycle, every 3 weeks for 3 cycles before radiation.
  Other Names: GEM
Drug: Cisplatin — Induction cisplatin 80mg/m2, every 3 weeks for 3 cycles before radiation; Concurrent cisplatin 100mg/m2, every 3 weeks for 2 cycles during radiation
  Other Names: DDP
Radiation: Intensity-modulated radiotherapy — Definitive intensity-modulated radiotherapy (IMRT) of 6996cGy will be given in 33 fractions.
  Other Names: IMRT

SUMMARY:
The trial aimed to compare cadonilimab combined with induction chemotherapy plus concurrent chemoradiotherapy (IC+CCRT) versus IC+CCRT alone in high-risk locoregionally-advanced nasopharyngeal carcinoma (LANPC).

DETAILED DESCRIPTION:
The trial plans to enroll patients with non-metastatic stage III-IVA (AJCC 8th, T4N1 or T1-4N2-3) locoregionally-advanced nasopharyngeal carcinoma (LANPC). Patients were randomly assigned in a 1:1 ratio to receive either gemcitabine-cisplatin induction chemotherapy and concurrent chemoradiotherapy (standard-therapy group) or cadonilimab combined with standard therapy (cadonilimab group). Cadonilimab was administered at a dosage of 10 mg per square meter intravenously once every 3 weeks for up to 17 cycles (3 induction cycles and 14 adjuvant cycles).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed nasopharyngeal carcinoma.
2. Tumor staged as III-IVA (AJCC 8th, except T3N0-1 or T4N0).
3. Eastern Cooperative Oncology Group performance status ≤1.
4. Adequate marrow function: neutrocyte count≥1.5×10e9/L, hemoglobin ≥90g/L and platelet count ≥100×10e9/L.
5. Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) ≤2.5×upper limit of normal (ULN), and bilirubin ≤ 1.5×ULN.
6. Adequate renal function: creatinine clearance rate ≥ 60 ml/min (Cockcroft-Gault formula).
7. Patients must be informed of the investigational nature of this study and give written informed consent.
8. Women of childbearing potential (WOCBP) who are sexually active must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of study drug. Men who are sexually active with WOCBP must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of the study drug

Exclusion Criteria:

1. Age > 65 or < 18.
2. Hepatitis B surface antigen (HBsAg) positive and hepatitis B virus DNA >1×10e3 copies/ml or 200IU/ml
3. Hepatitis C virus (HCV) antibody positive
4. Has active autoimmune disease, except type I diabetes, hypothyroidism treated with replacement therapy, and skin disease that doesn't require systemic treatment (e.g., vitiligo, psoriasis, or alopecia).
5. Has any condition that required systemic corticosteroid (equivalent to prednisone >10mg/d) or other immunosuppressive therapy within 28 days before informed consent. Patients received systemic corticosteroid equivalent to prednisone ≤10mg/d, inhale or topical corticosteroid will be allowed.
6. Has a known history of active TB (bacillus tuberculosis) within 1 year; patients with adequately treated active TB over 1 year ago will be allowed.
7. Has a known history of interstitial lung disease.
8. Has received a live vaccine within 30 days before informed consent or will receive a live vaccine in the near future.
9. Is pregnant or breastfeeding.
10. Prior malignancy within 5 years, except in situ cancer, adequately treated non-melanoma skin cancer, and papillary thyroid carcinoma.
11. Has known allergy to large molecule protein products or any compound of cadonilimab.
12. Has a known history of human immunodeficiency virus (HIV) infection.
13. Any other condition, including symptomatic heart failure, unstable angina, myocardial infarction, active infection requiring systemic therapy, mental illness or domestic/social factors, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interferes with the interpretation of the results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival (FFS) in intention-to-treat population | 3 years
  multiple endpoint 1: calculated from randomization to the date of locoregional recurrence, distant metastasis, or death from any cause, whichever occurred first.
Overall survival (OS) in intention-to-treat population | 3 years
  multiple endpoint 2: calculated from randomization to the date of death from any cause.

SECONDARY OUTCOMES:
Failure-free survival (FFS) in per-protocol population | 3 years
  calculated from randomization to the date of locoregional recurrence, distant metastasis, or death from any cause, whichever occurred first.
Overall survival (OS) in per-protocol population | 3 years
  calculated from randomization to the date of death from any cause.
Locoregional recurrence-free survival (LRRFS) | 3 years
  calculated from randomization to the date of locoregional persistence or 1st locoregional recurrence.
Distant metastasis-free survival (DMFS) | 3 years
  calculated from randomization to the date of first distant metastasis.
Adverse events (AEs) and serious adverse events (SAEs) | 3 years
  Graded according to CTCAE V5.0.
Quality of life (QoL) | week 1, 20, 40, 64
  The change of QoL from randomization to the start of radiotherapy, the end of radiotherapy, 13-16 weeks after radiotherapy, 2 years and 3 years after randomization. The EORTC QoL questionnaire-C30 (EORTC QLQ-C30）version 3.0 will be used. This questionnaire comprises 30 questions, 24 of which are aggregated into nine multi-question scales, that is, five functioning scales (e.g., physical), three symptom scales (e.g., fatigue) and one global health status scale. The remaining six single-question (e.g., dyspnoea) scales assess symptoms. These 15 scales will be scored according to the official Scoring Manual.
Failure-free survival (FFS) within different subgroups | 3 years
  analyses for FFS will be performed within the following subgroups: Epstein-Barr virus (EBV) DNA (≤4000copies/ml vs. >4000copies/ml), different PD-L1 expression levels, age, gender, performance status, T category, N category, and stage (III vs. IVA).
Tumor response | Through study completion, an average of 1.2 year
  Evaluation of tumor response as CR, PR, SD, PD, NA by clinicians

OTHER OUTCOMES:
Correlation between pre-treatment PD-L1 expression level and FFS | 3 years
  Pre-treatment PD-L1 expression level of tumor cell is evaluated centrally by means of immunohistochemical testing.
Evaluate failure-free survival in the subgroup of plasma Epstein-Barr virus DNA level | 3 years
  Subgroup analysis
Evaluate failure-free survival in the subgroup of clinical stage | 3 years
  Subgroup analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, M.D., Principal Investigator — Sun Yat-sen University
Locations (18):
- China (18):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Dongguan Peaple's Hospital, Dongguan, Guangdong
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Zhongshan city Peaple's Hospital, Zhongshan, Guangdong
  - Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Province Cancer Hosiptal, Wuhan, Hubei
  - Tongji Hospital Affiliated with Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital Affiliated with Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Shandong Province Cancer Hospital, Jinan, Shandong
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No
Complete de-identified patient data set will be submitted onto an online platform.

REFERENCES:
- [Result] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573
- [Result] Keam SJ. Cadonilimab: First Approval. Drugs. 2022 Aug;82(12):1333-1339. doi: 10.1007/s40265-022-01761-9. PMID 35986837
- [Result] Hsu C, Lee SH, Ejadi S, Even C, Cohen RB, Le Tourneau C, Mehnert JM, Algazi A, van Brummelen EMJ, Saraf S, Thanigaimani P, Cheng JD, Hansen AR. Safety and Antitumor Activity of Pembrolizumab in Patients With Programmed Death-Ligand 1-Positive Nasopharyngeal Carcinoma: Results of the KEYNOTE-028 Study. J Clin Oncol. 2017 Dec 20;35(36):4050-4056. doi: 10.1200/JCO.2017.73.3675. Epub 2017 Aug 24. PMID 28837405
- [Result] Ma BBY, Lim WT, Goh BC, Hui EP, Lo KW, Pettinger A, Foster NR, Riess JW, Agulnik M, Chang AYC, Chopra A, Kish JA, Chung CH, Adkins DR, Cullen KJ, Gitlitz BJ, Lim DW, To KF, Chan KCA, Lo YMD, King AD, Erlichman C, Yin J, Costello BA, Chan ATC. Antitumor Activity of Nivolumab in Recurrent and Metastatic Nasopharyngeal Carcinoma: An International, Multicenter Study of the Mayo Clinic Phase 2 Consortium (NCI-9742). J Clin Oncol. 2018 May 10;36(14):1412-1418. doi: 10.1200/JCO.2017.77.0388. Epub 2018 Mar 27. PMID 29584545